CLINICAL TRIAL: NCT00824005
Title: Randomized, Controlled, Phase II, Double-Blind Trial of Intramyocardial Injection of Autologous Bone Marrow Mononuclear Cells Under Electromechanical Guidance for Patients With Chronic Ischemic Heart Disease and Left Ventricular Dysfunction
Brief Title: Effectiveness of Stem Cell Treatment for Adults With Ischemic Cardiomyopathy (The FOCUS Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cardiovascular Cell Therapy Research Network (CCTRN) (Unknown)
Responsible Party: Principal Investigator, Dr Lemuel A Moye III, Professor - School of Public Health, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 580; U01HL087318 (NIH); 1 U01-HL-087318-01 (Project 3)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Ischemic Heart Disease; Left Ventricular Dysfunction; Angina; Ischemic Cardiomyopathy
Keywords: Congestive Heart Failure; Regional Wall Motion; Perfusion Defects
MeSH Terms: conditions — Ventricular Dysfunction, Left; Angina Pectoris; Heart Failure | interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Injections (Placebo Comparator): Participants will receive placebo injections.
  Interventions: Biological: Placebo
- Active Stem Cell Injections (Experimental): Participants will receive active stem cell injections.
  Interventions: Biological: Adult stem cells

INTERVENTIONS:
Biological: Adult stem cells — Single procedure of intramyocardial electromechanical-guided injection of approximately 100 million bone marrow mononucleated cells (BM-MNCs), administered in 15 different injection sites
  Other Names: Adult autologous stem cells; Bone marrow mononucleated cells
  Arms: Active Stem Cell Injections
Biological: Placebo — Single procedure of intramyocardial electromechanical-guided needle insertions and injection of 5% human serum albumin and saline in 15 different injection sites
  Other Names: Human serum albumin; HSA
  Arms: Placebo Injections

SUMMARY:
Coronary artery disease (CAD) is a common disorder that can lead to heart failure. Not all people with CAD are eligible for today's standard treatments. One new treatment approach uses stem cells-specialized cells capable of developing into other types of cells-to stimulate growth of new blood vessels for the heart. This study will determine the safety and effectiveness of withdrawing stem cells from someone's bone marrow and injecting those cells into the person's heart as a way of treating people with CAD and heart failure.

DETAILED DESCRIPTION:
Coronary artery disease (CAD), a disease in which blood vessels become clogged by a build-up of plaque, is the leading cause of heart failure, a condition in which the heart can no longer pump enough blood to the rest of the body. People with heart failure caused by CAD are said to have ischemic cardiomyopathy. Normal treatment for CAD involves coronary artery bypass grafting (in which a vein from another part of the body is grafted around an artery that has become blocked) or coronary angioplasty and stent placement (in which a blocked artery is opened and a small tube is placed to keep the artery open). However, some people with ischemic cardiomyopathy, such as those with substantial scar tissue on the heart wall or those with a particular heart structure, may not be eligible for these treatments. An alternative treatment being developed is therapeutic angiogenesis, which involves stimulating the growth of new blood vessels. Recent research has shown that withdrawing stem cells from bone marrow and implanting the cells into heart tissue may be an effective way to achieve therapeutic angiogenesis. This study will determine the safety and effectiveness of using stem cells to stimulate new blood vessel growth in the hearts of people with ischemic cardiomyopathy.

Participation in this study, including follow-up visits and phone calls, will last 60 months. Participants will first undergo 3 to 4 days of screening procedures that will include a physical examination, multiple lab tests, and a battery of tests on heart health. Next, participants will be randomized to receive either active stem cell injections or placebo injections. The injections and related procedures will be performed in a hospital and last approximately 72 hours. During this time, participants in both groups will first undergo a bone marrow aspiration procedure. Participants receiving active stem cells will also undergo NOGA electromechanical cardiac mapping, which involves inserting a monitoring device through a catheter and into the heart. Injections of stem cells will then be made to 15 damaged sites on the heart through a special catheter. Participants receiving placebo injections will receive 15 injections of an inactive, saline-based solution. After the injection procedures, all participants will undergo two echocardiograms, an electrocardiogram, blood tests, and overnight monitoring in a telemetry unit.

After the hospital stay, all participants will attend five study visits that will occur 1 week and 1, 3, 6, and 12 months after the injection procedures. At all study visits, participants will undergo an electrocardiogram, lab tests, and a review of adverse health events. On all but the last study visit, participants will have cardiac markers assessed, and they will wear a 24-hour Holter monitor to track heart activity. At the last three visits, participants will also complete quality of life questionnaires. All participants will then receive four follow-up telephone calls that will occur 2, 3, 4, and 5 years after the injection procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age with significant coronary heart disease not amenable to revascularization.
* Left ventricular dysfunction (LVEF) less than or equal to 45%, measured by echocardiogram; limiting angina (Class II to IV); and/or congestive heart failure (CHF), NYHA class II to III
* Receiving maximal medical therapy, defined as a medical regimen that includes the maximal tolerated dose of at least two antiangina medications, such as beta-blockers, nitrates, or calcium-channel blockers
* Presence of a defect, as identified by single photon emission computed tomography (SPECT) isotope protocol, or viability, as identified by NOGA electromechanical cardiac mapping system
* Coronary artery disease not well suited to any other type of revascularization procedure in the target region of the ventricle, as determined by a cardiovascular surgeon and interventional cardiologist who are not investigators in the trial
* Hemodynamic stability, as defined by systolic blood pressure of at least 80 mm Hg without intravenous pressors or support devices
* Females of childbearing potential must be willing to use two forms of birth control for the duration of the study

Exclusion Criteria:

* Atrial fibrillation or flutter without a pacemaker that guarantees a stable heart rate
* Unstable angina
* Left ventricular (LV) thrombus, as documented by echocardiography or LV angiography
* A vascular anatomy that precludes cardiac catheterization
* Severe valvular disease or mechanical aortic valve that precludes safe entry of the catheter into the left ventricle
* Pregnant or lactating
* Platelet count less than 100,000 per mm3
* White blood cell count less than 2,000 per mm3
* Revascularization within 30 days of consent
* Transient ischemic attack or stroke within 60 days of study consent
* Implantable cardioverter-defibrillator shock within 30 days of baseline consent, and within 30 days of randomization
* Presence of ventricular tachycardia lasting 30 seconds or more on 24-hour Holter monitor or electrocardiogram (ECG) performed during screening period
* Bleeding diathesis, defined as an international normalized ratio of at least 2.0 in the absence of warfarin therapy
* A history of malignancy in the last 5 years excluding basal cell carcinoma, that has been surgically removed, with proof of surgical clean margins
* Has a known history of HIV, has active hepatitis B or active hepatitis C
* Any condition requiring immunosuppressive medication
* High-risk acute coronary syndrome (ACS) or a myocardial infarction in the month prior to consent
* A left ventricular wall thickness of <8 mm (by echocardiogram) of the infero-lateral wall at the target site for cell injection.
* Inability to walk on a treadmill, except for class IV angina patients, who will be evaluated separately
* Enrolled in an investigational device or drug study within the previous 30 days
* Hepatic dysfunction, as defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 1.5 times the upper limit of normal range prior to study entry
* Chronic renal insufficiency, defined as a serum creatinine level greater than 2.5 mg/dL or requiring dialysis
* Any other condition that in the judgment of the investigator would be a contraindication to enrollment or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Simari, MD, Study Chair — Cardiovascular Cell Therapy Research Network
Locations (5):
- United States (5):
  - University of Florida-Department of Medicine, Gainesville, Florida
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Heart Institute, Houston, Texas

REFERENCES:
- [Background] Gee AP, Richman S, Durett A, McKenna D, Traverse J, Henry T, Fisk D, Pepine C, Bloom J, Willerson J, Prater K, Zhao D, Koc JR, Ellis S, Taylor D, Cogle C, Moye L, Simari R, Skarlatos S. Multicenter cell processing for cardiovascular regenerative medicine applications: the Cardiovascular Cell Therapy Research Network (CCTRN) experience. Cytotherapy. 2010 Sep;12(5):684-91. doi: 10.3109/14653249.2010.487900. PMID 20524773
- [Background] Willerson JT, Perin EC, Ellis SG, Pepine CJ, Henry TD, Zhao DX, Lai D, Penn MS, Byrne BJ, Silva G, Gee A, Traverse JH, Hatzopoulos AK, Forder JR, Martin D, Kronenberg M, Taylor DA, Cogle CR, Baraniuk S, Westbrook L, Sayre SL, Vojvodic RW, Gordon DJ, Skarlatos SI, Moye LA, Simari RD; Cardiovascular Cell Therapy Research Network (CCTRN). Intramyocardial injection of autologous bone marrow mononuclear cells for patients with chronic ischemic heart disease and left ventricular dysfunction (First Mononuclear Cells injected in the US [FOCUS]): Rationale and design. Am Heart J. 2010 Aug;160(2):215-23. doi: 10.1016/j.ahj.2010.03.029. PMID 20691824
- [Background] Zierold C, Carlson MA, Obodo UC, Wise E, Piazza VA, Meeks MW, Vojvodic RW, Baraniuk S, Henry TD, Gee AP, Ellis SG, Moye LA, Pepine CJ, Cogle CR, Taylor DA. Developing mechanistic insights into cardiovascular cell therapy: Cardiovascular Cell Therapy Research Network Biorepository Core Laboratory rationale. Am Heart J. 2011 Dec;162(6):973-80. doi: 10.1016/j.ahj.2011.05.024. PMID 22137069
- [Result] Perin EC, Willerson JT, Pepine CJ, Henry TD, Ellis SG, Zhao DX, Silva GV, Lai D, Thomas JD, Kronenberg MW, Martin AD, Anderson RD, Traverse JH, Penn MS, Anwaruddin S, Hatzopoulos AK, Gee AP, Taylor DA, Cogle CR, Smith D, Westbrook L, Chen J, Handberg E, Olson RE, Geither C, Bowman S, Francescon J, Baraniuk S, Piller LB, Simpson LM, Loghin C, Aguilar D, Richman S, Zierold C, Bettencourt J, Sayre SL, Vojvodic RW, Skarlatos SI, Gordon DJ, Ebert RF, Kwak M, Moye LA, Simari RD; Cardiovascular Cell Therapy Research Network (CCTRN). Effect of transendocardial delivery of autologous bone marrow mononuclear cells on functional capacity, left ventricular function, and perfusion in chronic heart failure: the FOCUS-CCTRN trial. JAMA. 2012 Apr 25;307(16):1717-26. doi: 10.1001/jama.2012.418. Epub 2012 Mar 24. PMID 22447880
- [Derived] Cogle CR, Wise E, Meacham AM, Zierold C, Traverse JH, Henry TD, Perin EC, Willerson JT, Ellis SG, Carlson M, Zhao DX, Bolli R, Cooke JP, Anwaruddin S, Bhatnagar A, da Graca Cabreira-Hansen M, Grant MB, Lai D, Moye L, Ebert RF, Olson RE, Sayre SL, Schulman IH, Bosse RC, Scott EW, Simari RD, Pepine CJ, Taylor DA; Cardiovascular Cell Therapy Research Network (CCTRN). Detailed analysis of bone marrow from patients with ischemic heart disease and left ventricular dysfunction: BM CD34, CD11b, and clonogenic capacity as biomarkers for clinical outcomes. Circ Res. 2014 Oct 24;115(10):867-74. doi: 10.1161/CIRCRESAHA.115.304353. Epub 2014 Aug 18. PMID 25136078
- See also: Click here for more information on the Cardiovascular Cell Therapy Research Network — http://www.cctrn.org
- See also: Click here for more information on the National Heart, Lung, and Blood Institute — http://www.nhlbi.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place at five Network centers and their associated satellite facilities between April 29, 2009 and April 18, 2011. The main centers are located in Ohio, Texas, Florida, Minnesota, and Tennessee. Study brochures, patient informational DVDs, and clinical trials.gov were among the tools used for recruitment.
Period: Overall Study
Arm/Group | Placebo Injections | Active Stem Cell Injections
Started | 31 | 61
Completed | 31 | 59
Not Completed | 0 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Injections | Active Stem Cell Injections | Total
Number analyzed (Participants) | 31 | 61 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.32 (8.25) | 63.95 (10.90) | 63.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 29 | 53 | 82
Region of Enrollment [Number; unit: participants]
  United States | 31 | 61 | 92

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximal Oxygen Consumption (VO2max)
Description: The VO2(max) is assessed using the Naughton treadmill protocol.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month VO2max data available are included.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Groups:
- Placebo Injections: Participants received placebo injections.
- Active Stem Cell Injections: Participants received active stem cell injections.
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 27 | 52
mL/kg/min | -0.6 (3.2) | 0.4 (2.8)
Statistical Analysis 1: Comparison: Placebo Injections vs Active Stem Cell Injections; Compare the change in the cell group to the change in the placebo group; Test type: Superiority or Other; p = 0.169, t-test, 2 sided — No adjustment for multiple comparisons; Mean Difference (Net) = 1.0, 95% CI 2-sided [-0.42 to 2.34], Standard Error of Mean 2.9

2. Primary Outcome: Change in Left Ventricular End Systolic Volume (LVESV)as Assessed Via Echo
Description: Echocardiographic measurements were performed by an echocardiographic core laboratory. LVESVs were calculated by the modified biplane Simpson method, using myocardial contrast to enhance endocardial definition. To account for patient body surface area, LVESV indices are reported.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and six month LVESV data available are included.
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 28 | 54
mL/m2 | 0 (10.8) | -0.9 (11.6)
Statistical Analysis 1: Comparison: Placebo Injections vs Active Stem Cell Injections; Change in the difference of end systolic volume over time; Test type: Superiority or Other; p = 0.856, t-test, 2 sided; Mean Difference (Net) = 1.0, 95% CI 2-sided [-10.05 to 12.07], Standard Error of Mean 23.9

3. Primary Outcome: Change in Reversible Defect Size
Description: Adenosine myocardial perfusion (SPECT) tests were collected at baseline and 6 months to identify change in ischemic (reversible) defects. SPECT imaging was performed at rest and after adenosine infusion over 4 minutes. To enhance the detection of viability on resting images, sublingual nitroglycerin was administered 15 minutes before injecting technetium Tc 99m sestamibi for the resting image.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and six month reversible defect data available are included.
Measure: Mean (Standard Deviation); unit: percentage of reversible defect
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 26 | 50
percentage of reversible defect | -2.7 (18.2) | -3.9 (25.4)
Statistical Analysis 1: Comparison: Placebo Injections vs Active Stem Cell Injections; Change in percent of the defect that is reversible; Test type: Superiority or Other; p = 0.835, t-test, 2 sided — Is the change in percent reversible defect the same between the two groups; Mean Difference (Net) = -1.2, 95% CI 2-sided [-12.5 to 10.1], Standard Error of Mean 22.3

4. Secondary Outcome: Regional Wall Motion by MRI (in Eligible Patients)
Description: Regional wall motion as measured by cardiac MRI (in patients who are not contraindicated)
Time Frame: Measured at Baseline and Month 6
Population: The small number of patients without contraindications for MRI (n=17) precluded performing informative analysis on the MRI data.
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Regional Blood Flow Improvement by MRI (in Eligible Patients)
Description: Regional blood flow improvement as measured by cardiac MRI (in patients who are not contraindicated)
Time Frame: Measured at Baseline and Month 6
Population: as for outcome 4
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Regional Wall Motion by Echocardiography
Description: Movement of the left ventricular wall measured in mm from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and six month wall motion data available are included.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 26 | 55
mm | 0 (0.4) | 0 (0.5)
Statistical Analysis 1: Comparison: Placebo Injections vs Active Stem Cell Injections; Difference in the change between the two groups; Test type: Superiority or Other; p = 0.471, t-test, 2 sided; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.30 to 0.14], Standard Error of Mean 0.5

7. Secondary Outcome: Clinical Improvement in CCS Classification (Angina Pectoris)
Description: Clinical improvement in Canadian Cardiovascular Society (CCS) functional classification of angina pectoris. The CCS scale ranges from Class I (best)"able to conduct ordinary daily activity without causing angina" to Class IV (worst) "Inability to perform any physical activity without discomfort; anginal symptoms may be present at rest." Patients receive a rating of 1-4 for their anginal symptoms. Results reflect the mean change in the total score over time.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and six month CCS data available are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 22 | 44
units on a scale | -0.3 (0.7) | -0.5 (0.8)
Statistical Analysis 1: Comparison: Placebo Injections vs Active Stem Cell Injections; Change in average improvement in Canadian Class Score over time between the two groups; Test type: Superiority or Other; p = 0.227, t-test, 2 sided; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.66 to 0.16], Standard Deviation 0.784

8. Secondary Outcome: Clinical Improvement in NYHA Classification
Description: Clinical improvement in New York Heart Association (NYHA) classification. The NYHA scale ranges from 1 (best)"Mild- no limitation of physical activity due to heart failure" to 4 (worst) "Severe-Unable to carry out any physical activity without discomfort due to heart failure". Patients receive a rating of 1-4 for their heart failure symptoms. Results reflect the mean change in the total score over time.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and six month NYHA class data available are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 30 | 55
units on a scale | -0.1 (0.7) | -0.3 (0.9)
Statistical Analysis 1: Comparison: Placebo Injections vs Active Stem Cell Injections; Difference in the change in NYHA score between the two groups; Test type: Superiority or Other; p = 0.361, t-test, 2 sided; Mean Difference (Net) = -0.176, 95% CI 2-sided [-0.56 to 0.21], Standard Error of Mean 0.845

9. Secondary Outcome: Number of Participants With a Decrease in Anti-anginal Medication
Description: Number of participants with a decrease in anti-anginal medication (nitrates needed weekly)
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and six month anti-anginal medication data available are included.
Measure: Number; unit: participants
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 28 | 50
participants | 0 | 2
Statistical Analysis 1: Comparison: Placebo Injections vs Active Stem Cell Injections; Difference in the change in anti-anginal meds across groups; Test type: Superiority or Other; p = 0.28, Chi-squared; Difference in the proportion of particip = 0.04, 95% CI 2-sided [-0.01 to 0.09], Standard Deviation 0.045

10. Secondary Outcome: Exercise Time and Level
Description: Exercise time and level as assessed via six minute walk test. (change in number of feet walked)
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and six month 6 minute walk data available are included.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 29 | 51
feet | 80 (415) | 184 (407)
Statistical Analysis 1: Comparison: Placebo Injections vs Active Stem Cell Injections; Change in six minute walk distance; Test type: Superiority or Other; p = 0.302, t-test, 2 sided; Mean Difference (Net) = 104, 95% CI 2-sided [-95 to 303], Standard Deviation 409

11. Secondary Outcome: Serum BNP Levels in Patients With CHF
Description: Serum b-type natriuretic peptide (BNP) levels in patients with congestive heart failure (CHF). A minority number of patients had pro-BNP collected versus regular BNP; these numbers are reported in the analysis population description.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and six month BNP data available are included.
Measure: Mean (Standard Deviation); unit: IUs
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 20 | 30
IUs
  BNP | 63 (249) | 28 (117)
  pro-BNP | 234 (1636) | 497 (1637)
Statistical Analysis 1: Comparison: Placebo Injections vs Active Stem Cell Injections; Difference in the change in BNP(reg) between cell and placebo group; Test type: Superiority or Other; p = 0.55, t-test, 2 sided; Mean Difference (Net) = -34.7, 95% CI 2-sided [-150 to 80], Standard Deviation 176

12. Secondary Outcome: LV Diastolic Dimension
Description: Left ventricular (LV) diastolic dimension as assessed by contrast echocardiography
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and six month LV diastolic data available are included.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 28 | 54
mL | -8.5 (34) | 0.9 (30)
Statistical Analysis 1: Comparison: Placebo Injections vs Active Stem Cell Injections; Change in the difference of end diastolic volume between the two groups over time; Test type: Superiority or Other; p = 0.198, t-test, 2 sided; Mean Difference (Net) = 9.5, 95% CI 2-sided [-5.03 to 23.93], Standard Deviation 31.2

13. Secondary Outcome: Incidence of a Major Adverse Cardiac Event
Description: Incidence of major adverse cardiac events (new MI, rehospitalization for PCI in coronary artery territories that were treated, death, or rehospitalization for acute coronary syndrome and for congestive heart failure).
  (Incidence rate)
Time Frame: Measured at Baseline and Month 6
Population: Incidence of major adverse cardiac events between baseline and 6 months. (Incidence rate)
Measure: Number; unit: events
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 31 | 61
events | 4 | 5
Statistical Analysis 1: Comparison: Placebo Injections vs Active Stem Cell Injections; The difference in the incidence of major adverse cardiac events between the two groups over time. (Incidence rate); Test type: Superiority or Other; p = 0.47, t-test, 2 sided; Difference in the incidence rates = -0.047, 95% CI 2-sided [-0.133 to 0.039], Standard Error of Mean 0.044

14. Secondary Outcome: Reduction in Fixed Perfusion Defect(s)Via SPECT
Description: Fixed total defect is the stress total defect minus the reversible component.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and six month fixed defect data available are included.
Measure: Mean (Standard Deviation); unit: percentage of defect that is fixed
Arm/Group | Placebo Injections | Active Stem Cell Injections
Number analyzed (Participants) | 25 | 52
percentage of defect that is fixed | 1.9 (7.7) | 1.2 (8.7)
Statistical Analysis 1: Comparison: Placebo Injections vs Active Stem Cell Injections; Difference in the change between the two groups; Test type: Superiority or Other; p = 0.7, t-test, 2 sided; Mean Difference (Net) = -0.7, 95% CI 2-sided [-4.78 to 3.36], Standard Error of Mean 8.4

ADVERSE EVENTS:
Time Frame: Events reported are from Randomization Date to the 6 month endpoint data collection window (i.e. 210 days post intervention)
Arm/Group | Placebo Injections | Active Stem Cell Injections
Serious Adverse Events (participants affected / at risk) | 6/31 | 9/61
Other Adverse Events (participants affected / at risk) | 11/31 | 19/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Injections (N=31) | Active Stem Cell Injections (N=61)
Chest pain (Cardiac disorders) | 2 (3) | 4 (4)
Tachycardia (Cardiac disorders) | 1 (1) | 3 (7)
Heart Failure (Cardiac disorders) | 3 (5) | 2 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Injections (N=31) | Active Stem Cell Injections (N=61)
Tachycardia (Cardiac disorders) | 3 (3) | 3 (5) — Tachycardia not requiring hospitalization or a change to current therapy
Nausea (Gastrointestinal disorders) | 2 (4) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Change in BNP levels (Cardiac disorders) | 3 (3) | 8 (8)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
Sample size was small and required large improvements in order to show significant treatment effects. SPECT often underestimates reversibility and viability in those with multivessel disease. Presence of cardiac devices limited MRI evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes